CLINICAL TRIAL: NCT01387542
Title: An Open-label, PRospective Study to Evaluate Social Function and Overall Improvement of Paliperidone ER Treatment in Thai Schizophrenia PatieNT (PRESENT)
Brief Title: Safety and Efficacy Study of Paliperidone Extended Release (ER) Among Thai Schizophrenia Participants
Acronym: PRESENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015976; R076477SCH4037 (Other: Janssen-Cilag Ltd.,Thailand)
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Extended Release (ER); INVEGA
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Extended Release (ER) (Experimental): Paliperidone ER 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral tablets depending on investigator's discretion once daily for 10 weeks
  Interventions: Drug: Paliperidone extended release (ER)

INTERVENTIONS:
Drug: Paliperidone extended release (ER) — Paliperidone ER 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral tablets depending on investigator's discretion once daily for 10 weeks

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of paliperidone extended release (ER) treatment in Thai schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), non-randomized (the study drug is not assigned by chance) study to evaluate the efficacy and safety of paliperidone ER in adult Thai schizophrenia participants. The study consists of a screening phase and an open-label treatment phase. Study duration will be 10 weeks and participants can either be inpatient or outpatient. The recommended paliperidone ER starting and maintenance dose will be 6 milligram (mg) per day for most participants. Throughout the study, flexible dosing ranging from 3 to 12 mg per day may be used at the discretion of the investigator. Throughout the study, participants will be evaluated for efficacy using clinician rating (Clinical and Global Impressions-Severity [CGI-S] scale, and Personal and Social Performance Scale [PSP]) scales. Safety of the participants will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self)
* Participants unsatisfied with their previous treatment
* Previously or currently on oral atypical antipsychotics

Exclusion Criteria:

* Serious unstable medical condition, including recent and present clinically relevant laboratory abnormalities
* History or current symptoms of tardive dyskinesia (twitching or jerking movements that you cannot control in your face, tongue, or other parts of your body)
* History of neuroleptic malignant syndrome (high fever, rigid muscles, shaking, confusion, sweating more than usual, increased heart rate or blood pressure, or muscle pain or weakness)
* Pregnant or breast-feeding female
* Participation in an investigational drug trial within 30 days prior to selection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (2):
- Thailand (2):
  - Chiang Mai
  - Songkhla

REFERENCES:
- See also: An Open-label, PRospective Study to Evaluate Social Function and Overall Improvement of Paliperidone ER Treatment in Thai Schizophrenia PatieNT (PRESENT) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1106&filename=CR015976_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER)
Started | 40
Treated | 38
Completed | 32
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Changed diagnosis | 1
Not completed — Insufficient response | 1
Not completed — Non-compliant | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.13 (12.314)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale at Week 10
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening .
Time Frame: Baseline, Week 10
Population: Intent-To-Treat (ITT) population included participants who received at least 1 dose of study medication and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 38
Units on a scale
  Baseline | 3.55 (1.155)
  Change at Week 10 | 0.82 (1.036)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER); Test type: Superiority or Other; p = 0.000, Friedman test

2. Primary Outcome: Change From Baseline in Personal and Social Performance (PSP) Total Score at Week 2
Description: The PSP scale assesses degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Score ranges from 1 to 100, divided into 10 equal intervals to rate degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Based on 4 domains there will be 1 total score. Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline, Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 38
Units on a scale
  Baseline | 58.95 (15.710)
  Change at Week 2 | -4.289 (9.647)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER); Test type: Superiority or Other; p = 0.009, Paired t-test

3. Primary Outcome: Change From Baseline in Personal and Social Performance (PSP) Total Score at Week 6
Description: as for outcome 2
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 38
Units on a scale | -7.053 (11.463)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER); Test type: Superiority or Other; p = 0.001, Paired t-test

4. Primary Outcome: Change From Baseline in Personal and Social Performance (PSP) Total Score at Week 10
Description: as for outcome 2
Time Frame: Baseline, Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 38
Units on a scale | -9.868 (14.640)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER); Test type: Superiority or Other; p = 0.000, Paired t-test

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Paliperidone Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 22/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone Extended Release (ER) (N=40)
Mania (Psychiatric disorders) | 1 (1)
Elevated mood (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=40)
Drowsiness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 5
Extrapyramidal disorder (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Hypotension (Vascular disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 2
Palpitation (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2

LIMITATIONS AND CAVEATS:
Study had an open-label trial design with lack of a comparator arm; therefore it was difficult to conclude the efficacy and safety results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review results communications prior to publication and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The paper that incorporates confidential information requires Sponsor's written consent. PI will withhold publication for up to an additional 60 days to allow for filing of a patent application.